CLINICAL TRIAL: NCT04405843
Title: Randomized, Placebo Controlled, Double Blind Clinical Trial to Evaluate the Efficacy of Molecule D11AX22 in Adults Patients From Valle Del Cauca, Colombia With Early Stages of SARS COV2 / COVID-19
Brief Title: Efficacy of Ivermectin in Adult Patients With Early Stages of COVID-19 (EPIC Trial)
Acronym: EPIC
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centro de Estudios en Infectogía Pediatrica (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ScDi823; IVE-PA (Other: INVIMA (Colombian Regulatory Agency))
Record Dates: First submitted 2020-05-23; First posted 2020-05-28 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2020-12

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Ivermectin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ivermectin (Experimental): Ivermectin, 300 micrograms / kg, once daily for 5 days
  Interventions: Drug: Ivermectin Oral Product
- Placebo (Placebo Comparator): Substance with similar physical and organoleptic characteristics as ivermectin, without the active drug ingredient
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ivermectin Oral Product — Ivermectin oral suspension, 6 mg/mL
  Arms: Ivermectin
Drug: Placebo — Substance with similar physical and organoleptic characteristics as ivermectin, without the active drug ingredient
  Arms: Placebo

SUMMARY:
Double blind, placebo controlled, randomized clinical trial to evaluate the efficacy of ivermectin in preventing progression of disease in adult patients with early stages of COVID-19

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Confirmed SARS-CoV-2 by RT-PCR or antigen detection in a Colombian NIH-approved laboratory
* Beginning of symptoms in the past 7 days
* Mild disease
* Informed consent

Exclusion Criteria:

* Preexisting liver disease
* Hypersensitivity to ivermectin
* Participants in other clinical trials for therapies against COVID-19
* Severe pneumonia
* Pregnant or breastfeeding women
* Concomitant use of warfarin, erdafitinib or quinidine
* Use of ivermectin in the 5 days prior to randomization
* Inability to obtain a blood sample needed to assess liver transaminases
* Elevation of transaminases >1.5 times the normal level
* Participant whose first contact with the study personnel occurs between days 5 and 7 and at that time manifests significant and progressive resolution of COVID-19 related signs and symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 476 (Actual)
Dates: Start 2020-07-14 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2020-12-21 (Actual)

PRIMARY OUTCOMES:
Time to event | 21 days
  Time until resolution of symptoms

SECONDARY OUTCOMES:
Clinical condition on day 2 | On day 2 (± 1 day) after randomization
  Clinical condition in an ordinal scale of 7 points, on day 2. Higher scores indicate worse outcomes
Clinical condition on day 5 | On day 5 (± 1 day) after randomization
  Clinical condition in an ordinal scale of 7 points, on day 5. Higher scores indicate worse outcomes
Clinical condition on day 8 | On day 8 (± 1 day) after randomization
  Clinical condition in an ordinal scale of 7 points, on day 8. Higher scores indicate worse outcomes
Clinical condition on day 11 | On day 11 (± 1 day) after randomization
  Clinical condition in an ordinal scale of 7 points, on day 11. Higher scores indicate worse outcomes
Clinical condition on day 15 | On day 15 (± 1 day) after randomization
  Clinical condition in an ordinal scale of 7 points, on day 15. Higher scores indicate worse outcomes
Clinical condition on day 21 | On day 21 (± 1 day) after randomization
  Clinical condition in an ordinal scale of 7 points, on day 21. Higher scores indicate worse outcomes
Proportion of subjects with additional care | 21 days
  Proportion of subjects who require hospitalization, use of supplementary oxygen for >24 hours or ICU admission
Proportion of subjects who die | From randomization up to 21 days
  Proportion of subjects who die
Duration of additional care | 21 days
  Duration of supplementary oxygen, hospitalization, ICU stay
Adverse events | 21 days
  Proportion of subjects who develop solicited adverse events
Proportion of subjects who discontinue intervention | 21 days
  Proportion of subjects who required discontinuation of the intervention due to adverse events
Time to event | 21 days
  Time until deterioration of 2 or more points in an ordinal 7 points scale.
Duration of fever | 21 days
  Number of days with fever since randomization

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo López-Medina, MD MSc, Principal Investigator — Scientific Director of Centro de Estudios en Infectología Pediátrica --CEIP--
Locations (1):
- Centro de Estudios en Infectología Pediátrica, Cali, Valle del Cauca Department, Colombia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Derived] Lopez-Medina E, Lopez P, Hurtado IC, Davalos DM, Ramirez O, Martinez E, Diazgranados JA, Onate JM, Chavarriaga H, Herrera S, Parra B, Libreros G, Jaramillo R, Avendano AC, Toro DF, Torres M, Lesmes MC, Rios CA, Caicedo I. Effect of Ivermectin on Time to Resolution of Symptoms Among Adults With Mild COVID-19: A Randomized Clinical Trial. JAMA. 2021 Apr 13;325(14):1426-1435. doi: 10.1001/jama.2021.3071. PMID 33662102